CLINICAL TRIAL: NCT07209982
Title: Dual Task Training Versus Single Task Training in Chronic Hemiplegic Stroke Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lahore (Other)
Responsible Party: Principal Investigator, Rabiya Sadaf, Student, University of Lahore
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UOL/IREB/25/09/0048
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Hemiplegia; Hemiplegia Following Ischemic Stroke; Stroke
Keywords: Balance; Dual-task training; Gait; Hemiplegic stroke; Rehablitation
MeSH Terms: conditions — Hemiplegia; Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual-Task Training (DTT) (Experimental): Participants receive structured gait and balance training combined with a concurrent secondary task. Secondary tasks include simple cognitive challenges (such as counting backward or naming objects) or light motor tasks (such as carrying a cup or tossing a ball). Sessions are 60 minutes, three times per week for six weeks, delivered under therapist supervision. Task difficulty is gradually increased while maintaining safety.
  Interventions: Behavioral: Dual-Task Training (DTT)
- Single-Task Training (STT) (Active Comparator): Participants receive the same dose of gait and balance training as the experimental arm, but without any concurrent secondary task. Exercises include level walking, directional changes, obstacle negotiation, and balance tasks on stable or unstable surfaces. Sessions are 60 minutes, three times per week for six weeks, supervised by a therapist. Difficulty is progressed through physical task demands only.
  Interventions: Behavioral: Single-Task Training (STT)

INTERVENTIONS:
Behavioral: Dual-Task Training (DTT) — This intervention combines gait and balance practice with a simultaneous secondary task to mimic real-world multitasking demands. Participants complete 60-minute sessions, three times per week for six weeks. Secondary tasks include simple cognitive activities (such as serial subtraction, word recall, or visual scanning) or light motor tasks (such as carrying an object or tossing a ball). Task complexity is increased gradually according to participant tolerance. All sessions are supervised by a trained physiotherapist, with rest breaks and safety precautions provided.
  Other Names: Cognitive-Motor Dual-Task Training (CMDT)
  Arms: Dual-Task Training (DTT)
Behavioral: Single-Task Training (STT) — This intervention provides gait and balance training without any added secondary tasks. Participants complete 60-minute sessions, three times per week for six weeks. Exercises include level walking, directional changes, obstacle negotiation, static and dynamic balance activities, and surface progressions (such as standing on foam). Progression is achieved by altering the physical task difficulty only. Sessions are supervised by a physiotherapist with safety measures in place and rest breaks as needed.
  Arms: Single-Task Training (STT)

SUMMARY:
What is this study about? This study compares two common ways of practicing walking and balance after a stroke: (1) dual-task training, where a person walks or balances while doing a second task (such as counting backward or carrying a light object), and (2) single-task training, where a person practices walking and balance without any extra task. The goal is to learn whether practicing with or without an added task is more practical and acceptable for people living with long-standing weakness on one side of the body (hemiplegia) after stroke.

Why is this important? Many everyday activities-walking while talking, looking for a bus, or carrying a bag-require attention to more than one thing at a time. Some stroke survivors find this difficult. Training that safely mimics real-life multitasking may help therapists design better rehabilitation plans.

Who can take part? Adults aged 45-65 years with a diagnosis of hemiplegic stroke who can walk without hands-on help may be eligible. People with other neurological conditions that affect walking, severe problems with understanding or communication, or recent serious medical/surgical issues will not be included. Additional screening will check safety for exercise.

What will happen if I join?

Participants are randomly assigned (like a coin toss) to one of two groups:

Dual-task training group: walking/balance activities plus a simple cognitive or motor task.

Single-task training group: the same walking/balance activities without any extra task.

Both groups attend 60-minute sessions, three times per week, for six weeks at The University of Lahore Teaching Hospital or Sehat Medical Complex. A trained therapist supervises all sessions and adjusts difficulty gradually. Short rest breaks are provided.

What will be measured? At baseline, 2 weeks, 4 weeks, and 6 weeks, an assessor who does not know the assigned group will record walking and balance using the Tinetti Performance-Oriented Mobility Assessment (POMA). Safety (such as any falls, dizziness, or discomfort) and attendance will also be recorded.

What are the possible risks and benefits? Risks are similar to supervised physiotherapy: temporary muscle soreness, fatigue, or loss of balance. Therapists use safety measures (close supervision, stable equipment, and rest periods). Participants may experience the general benefits of structured rehabilitation (practice, education, and monitored activity). Taking part is voluntary, and usual care remains available.

Privacy and cost Personal information is kept confidential and stored securely. There is no payment for participation. There are no charges for study-related therapy sessions.

Time commitment About 18 sessions over 6 weeks, plus four short assessment visits.

Contacts Study team members can answer questions at any time and will obtain written informed consent before any study procedures begin.

DETAILED DESCRIPTION:
Study design and setting Single-center, parallel-group, randomized, single-blind controlled trial conducted at the University Institute of Physical Therapy (UIPT), Faculty of Allied Health Sciences, The University of Lahore, with sessions delivered at the University of Lahore Teaching Hospital and Sehat Medical Complex.

Rationale After stroke, many individuals report difficulty walking when attention is divided. Rehabilitation programs often use either single-task practice or add a concurrent cognitive or motor task to approximate everyday demands. A standardized comparison of these two approaches over a fixed dose of therapy can inform practical rehabilitation planning.

Participants

Target population: Adults (45-65 years) with hemiplegic stroke who can ambulate without physical assistance.

Key inclusion criteria: clinical diagnosis of hemiplegic stroke; able to follow instructions; ambulatory (with or without an assistive device but without hands-on help).

Key exclusion criteria: other neurological conditions affecting mobility; severe cognitive-communication impairment that prevents following instructions; recent acute medical or surgical conditions that make exercise unsafe; severe hemiparesis that prevents safe participation.

Eligibility is confirmed by screening interview and brief clinical examination.

Sample size and allocation Planned enrollment is 62 participants, randomized 1:1 to dual-task training (DTT) or single-task training (STT). Randomization uses sequentially numbered, opaque, sealed envelopes prepared by an investigator not involved in treatment or assessments. Group assignment is concealed until after baseline testing.

Blinding Outcome assessments are conducted by a trained assessor blinded to group allocation. Due to the nature of exercise interventions, therapists and participants are not blinded.

Interventions (dose matched) All sessions last 60 minutes, 3 times per week for 6 weeks (approximately 18 total sessions). Sessions include a brief warm-up, progressive task practice, and short rest breaks. Safety measures include therapist supervision, use of gait belts where appropriate, and removal of environmental hazards.

Dual-task training (DTT):

Gait tasks: level walking, directional changes, obstacle negotiation, and surface progressions (e.g., foam).

Concurrent tasks: simple cognitive tasks (e.g., counting backward by ones or threes; identifying targets in the environment; short memory queries) or light motor tasks (e.g., carrying a half-filled cup; gentle ball toss).

Progression: Gradual increase in task complexity (e.g., longer walking paths, slightly more challenging arithmetic, modestly increased obstacle height) while maintaining safety and allowing rest.

Single-task training (STT):

Gait tasks: matched to DTT (level walking, directional changes, obstacle negotiation, surface progressions) without any concurrent cognitive or secondary motor task.

Balance tasks: static and dynamic balance (single-leg stance as able; reaching tasks; stance on foam; graded perturbation practice) without any added task.

Progression: Similar physical progression as DTT (e.g., speed, distance, surface challenge) with therapist supervision.

Outcome measures and schedule

Assessments occur at Baseline, Week 2, Week 4, and Week 6:

Primary outcomes:

Tinetti Performance-Oriented Mobility Assessment (POMA) - Balance subscore (0-16) and Gait subscore (0-12).

Process and safety monitoring: session attendance, adverse events (falls, near-falls, dizziness, pain), and participant-reported fatigue during therapy.

The assessor records scores using standardized instructions. To minimize bias, participants are asked not to reveal their group to the assessor.

Visit structure

Screening/Baseline visit (about 45-60 minutes): informed consent; eligibility check; demographics; baseline POMA testing; safety counseling.

Treatment visits (60 minutes each): warm-up, structured task practice per group, monitored rest breaks, cool-down, safety check.

Interim assessments (Week 2 and Week 4; 15-30 minutes): POMA testing by the blinded assessor.

End-of-program assessment (Week 6; 30-45 minutes): final POMA testing; safety review; discussion of next-step clinical follow-up outside the study as needed.

Safety measures Therapists supervise all activities, provide guarding for balance tasks, and adapt difficulty based on participant tolerance. Any adverse events are documented and reported per institutional policy. Participants may pause or stop a session at any time.

Data management and confidentiality Paper forms and electronic records are stored securely with restricted access. Study data are coded; identifying information is kept separate from outcome data. Only authorized team members may access the linkage file. Data will be analyzed in aggregate without naming individuals.

Participant rights Participation is voluntary. Individuals may decline or withdraw at any time without affecting their access to usual care. There is no financial cost for study-related sessions. Transportation and scheduling needs are accommodated as feasible.

Training fidelity Intervention checklists specify the planned activities and progression for each week to ensure comparable dose and content across therapists and participants. Periodic supervision verifies adherence to the protocol.

Dissemination plan Findings from this protocol will be shared in academic venues and with local rehabilitation teams in a way that protects participant privacy. Individual results are not reported; only grouped, de-identified data are shared.

Contacts For questions about the study procedures, eligibility, scheduling, or privacy, potential participants and healthcare providers may contact the study team at the University Institute of Physical Therapy, The University of Lahore. Written informed consent will be obtained before any study-specific activities begin.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemiplegic stroke (Nam, 2023)
* Both males and females patients
* Participants ≤ 6 months poststroke (Nam, 2023)
* Participants age between 45-65(Zhou et al., 2021)
* Patients who are able to walk without assistance.(Joya, 2023) .

Exclusion Criteria:

* History of other neurological conditions effecting mobility (Muzio et al., 2023).
* Severe cognitive impairments or communication difficulties. (Liu et al., 2017)
* Recent acute medical/surgical conditions unrelated to stroke.(Nam, 2023)
* Other Systemic disease
* Participants with severe hemiparesis who are unable to produce movement accurately (Zhang et al., 2022).

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-08-19 (Actual); Study Completion 2025-09-24 (Actual)

PRIMARY OUTCOMES:
Change in Balance Performance (Tinetti Balance Subscore) | Baseline, 2 weeks, 4 weeks, and 6 weeks
  The balance component of the Tinetti Performance-Oriented Mobility Assessment (POMA), scored 0-16, with higher scores indicating better balance. Used to evaluate static and dynamic balance during standing and transitional tasks.
Change in Gait Performance (Tinetti Gait Subscore) | Baseline, 2 weeks, 4 weeks, and 6 weeks
  The gait component of the Tinetti POMA, scored 0-12, assessing step length, symmetry, initiation, path deviation, and trunk stability during walking. Higher scores indicate better gait performance.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Lahore Teaching Hospital, Lahore, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pang MYC, Yang L, Ouyang H, Lam FMH, Huang M, Jehu DA. Dual-Task Exercise Reduces Cognitive-Motor Interference in Walking and Falls After Stroke. Stroke. 2018 Dec;49(12):2990-2998. doi: 10.1161/STROKEAHA.118.022157. PMID 30571419